CLINICAL TRIAL: NCT02848703
Title: Study " COFLORES ":Imaging of Coronary Reserve Without Tracers
Brief Title: Study " COFLORES "
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-45; 2016-A00026-45 (Registry Identifier: ansm)
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Perfusion
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Device: Magnetic Resonance Imaging (MRI); Device: phosphorus-31 Magnetic Resonance Spectroscopy; Device: sodium-23 MRI

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI)
Device: phosphorus-31 Magnetic Resonance Spectroscopy
Device: sodium-23 MRI

SUMMARY:
Myocardial perfusion is a major parameter characterizing the status of capillary circulation of the myocardium. Its quantification is possible using Magnetic Resonance Imaging (MRI) during the 1st pass of a contrast agent through the capillary system. This technique is radiation-free, but it is difficult to repeat measurements during a single exam. Also, a number of patients suffering from cardiac disease cannot receive contrast agent injections. The investigators have developed a totally non-invasive approach for quantifying myocardial perfusion. It is based on the magnetic labeling of arterial spins. Flowing into the capillaries (Arterial spin labeling, ASL).

Goal : The major goal of this research protocol is to validate a totally non-invasive method of myocardial blood flow quantification using MRI without contrast agent injection

ELIGIBILITY:
Inclusion Criteria:

* People having no heart disease or treatment referred to cardiology
* People having no cons -indications to MRI
* People having no cons -indications to gadolinium ;
* People not wearing implantable devices
* People not wearing metallic foreign bodies or risk (eg . Business of steel, etc .. )
* People having no cardiovascular risk factor
* Person subject to the social security scheme
* Nobody agreeing to participate in the study and who signed the informed consent

Exclusion Criteria:

* Refusal to go spontaneous or MRI because of claustrophobia important
* Trouble rhythm making MRI uninterpretable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion | 1day
  MRI based on the magnetic labeling of arterial spins

SECONDARY OUTCOMES:
the myocardial energetic status | 1day
  using phosphorus-31 Magnetic Resonance Spectroscopy
the myocardial sodium | 1day
  using sodium-23 MRI

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No